CLINICAL TRIAL: NCT04959032
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Lumateperone for the Prevention of Relapse in Patients With Schizophrenia
Brief Title: Lumateperone for the Prevention of Relapse in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-304
Record Dates: First submitted 2021-06-30; First posted 2021-07-12 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Relapse Prevention; Maintenance Design
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone 42 mg (Experimental)
  Interventions: Drug: Lumateperone 42 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumateperone 42 mg — Lumateperone 42 mg capsules administered orally, once daily.
  Arms: Lumateperone 42 mg
Drug: Placebo — Matching capsules administered orally, once daily.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, fixed-dose study in adult patients with a primary diagnosis of schizophrenia according to criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, (DSM-5).

DETAILED DESCRIPTION:
The study will be conducted in the following 5 phases:

* A no-drug Screening Phase up to 7 days in duration during which patient eligibility will be assessed;
* A 6-week, open-label Run-in Phase (RIP) during which all patients will receive oral lumateperone 42 mg/day;
* A 12-week, open-label Stabilization Phase (SP) during which all patients will receive oral lumateperone 42 mg/day;
* A Double-blind Treatment Phase (DBTP) 26 weeks in duration during which patients receive either lumateperone 42 mg or placebo (1:1 ratio);
* A 2-week Safety Follow-up (SFU) Phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 60 years of age, inclusive.
* Current diagnosis of schizophrenia according to DSM-5 criteria as determined by the modified Structured Clinical Interview for DSM-5 (modified SCID-5).
* Diagnosis of schizophrenia for a minimum of 1 year before Visit 1.
* Current psychotic episode < 4 weeks duration at Visit 1.
* PANSS total score ≥ 70 and ≤ 120 at Visit 1 and Visit 2.
* Rating of at least 4 (moderate) on at least two of the following four PANSS positive symptoms: delusions (P1), hallucinatory behavior (P3), conceptual disorganization (P2), suspiciousness/persecution (P6) at Visit 1 and Visit 2.
* Patient must identify a caregiver who provides consents to participate in the study.
* In the opinion of the Investigator, the patient has significant risk for suicidal behavior during the course of his/her participation in the study.

Exclusion Criteria:

* Currently meeting DSM-5 criteria for any of the following:

Schizoaffective disorder, schizophreniform disorder, and other psychotic disorders; Bipolar I or Bipolar II Disorder; Intellectual developmental disorder, delirium, dementia, amnestic and other cognitive disorders; Known or suspected borderline or antisocial personality disorder or other DSM 5 personality disorder of sufficient severity to interfere with participation in this study; Substance use disorder (other than nicotine) within the 3 months prior to Visit 1 of this study.

* Patients in their first episode of psychosis.
* Treatment-resistant schizophrenia over the last 2 years, defined as little or no symptomatic response to at least 2 courses of antipsychotic treatment of an adequate duration (at least 6 weeks) and at a therapeutic dose (according to the package insert for the antipsychotic treatment).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Time to first symptom relapse during the Double-blind Treatment Phase | Number of days from the randomization date to the first relapse date up to 26 weeks.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (21):
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Bellflower, California
  - Clinical Site, Cerritos, California
  - Clinical Site, Culver City, California
  - Clinical Site, Garden Grove, California
  - Clinical Site, Lemon Grove, California
  - Clinical Site, Montclair, California
  - Clinical Site, Orange, California
  - Clinical Site, Hollywood, Florida
  - Clinical Site, Miami Lakes, Florida
  - Clinical Site, Oakland Park, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Las Vegas, Nevada
  - Clinical Site, Berlin, New Jersey
  - Clinical Site, North Canton, Ohio
  - Clinical Site, Austin, Texas
  - Clinical Site, DeSoto, Texas
  - Clinical Site, Richardson, Texas
- Bulgaria (14):
  - Clinical Site, Burgas
  - Clinical Site, Kardzhali
  - Clinical Site, Kazanlak
  - Clinical Site, Lovech
  - Clinical Site, Novi Iskar
  - Clinical Site, Pleven
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Targovishte
  - Clinical Site, Tsarev Brod
  - Clinical Site, Tserova Koria
  - Clinical Site, Veliko Tarnovo
  - Clinical Site, Vratsa
- Poland (3):
  - Clinical Site, Gdansk
  - Clinical Site, Gorlice
  - Clinical Site, Tuszyn
- Serbia (4):
  - Clinical site, Belgrade
  - Clinical Site, Kovin
  - Clinical Site, Kragujevac
  - Clinical Site, Novi Kneževac

IPD SHARING:
Plan to Share IPD: No